CLINICAL TRIAL: NCT02464449
Title: Patient-Centered Pain Care Using Artificial Intelligence and Mobile Health Tools
Acronym: REACT (AI CBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 13-350
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Back Pain
Keywords: Cognitive Behavioral Therapy; Mobile Health Technology; Patient Care Management
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI CBT (Experimental): AI CBT engine will make recommendations to step-down or step-up intensity of CBT FU based on what patient reports and what other similar patients report. Stepped care model.
  Interventions: Behavioral: Behavioral: AI-CBT
- Standard telephone CBT (Active Comparator): Controls receive 10 hour-long standard telephone CBT sessions, a pedometer/log after baseline, and a Patient Handbook.
  Interventions: Behavioral: Behavioral: Standard Telephone CBT

INTERVENTIONS:
Behavioral: Behavioral: AI-CBT — AI CBT engine will make recommendations to step-down or step-up intensity of CBT follow-up based on what patient reports and what other similar patients report. Stepped care model.
  Arms: AI CBT
Behavioral: Behavioral: Standard Telephone CBT — Controls receive 10 hour-long standard telephone CBT sessions, a pedometer/log after baseline, and a Patient Handbook.
  Arms: Standard telephone CBT

SUMMARY:
This study will evaluate a new approach for back pain care management using artificial intelligence and evidence-based cognitive behavioral therapy (AI-CBT) so that services automatically adapt to each Veteran's unique needs, achieving outcomes as good as standard care but with less clinician time.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) is one of the most effective treatments for chronic back pain. However, only half of Veterans have access to trained CBT therapists, and program expansion is costly. Moreover, VA CBT programs consist of 10 weekly hour-long sessions delivered using an approach that is out-of-sync with stepped-care models designed to ensure that scarce resources are used as effectively and efficiently as possible. Data from prior CBT trials have documented substantial variation in patients' needs for extended treatment, and the characteristics of effective programs vary significantly. Some patients improve after the first few sessions while others need more extensive contact. After initially establishing a behavioral plan, still other Veterans may be able to reach behavioral and symptom goals using a personalized combination of manuals, shorter follow-up contacts with a therapist, and automated telephone monitoring and self-care support calls. In partnership with the National Pain Management Program, the investigators propose to apply state-of-the-art principles from "reinforcement learning" (a field of artificial intelligence or AI used successfully in robotics and on-line consumer targeting) to develop an evidence-based, personalized CBT pain management service that automatically adapts to each Veteran's unique and changing needs (AI-CBT). AI-CBT will use feedback from patients about their progress in pain-related functioning measured daily via pedometer step-counts to automatically personalize the intensity and type of patient support; thereby ensuring that scarce therapist resources are used as efficiently as possible and potentially allowing programs with fixed budgets to serve many more Veterans. The specific aims of the study are to: (1) demonstrate that AI-CBT has non-inferior pain-related outcomes compared to standard telephone CBT; (2) document that AI-CBT achieves these outcomes with more efficient use of scarce clinician resources as evidenced by less overall therapist time and no increase in the use of other VA health services; and (3) demonstrate the intervention's impact on proximal outcomes associated with treatment response, including program engagement, pain management skill acquisition, satisfaction with care, and patients' likelihood of dropout. The investigators will use qualitative interviews with patients, clinicians, and VA operational partners to ensure that the service has features that maximize scalability, broad scale adoption, and impact. 278 patients with chronic back pain will be recruited from the VA Connecticut Healthcare System and the VA Ann Arbor Healthcare System, and randomized to standard 10-sessions of telephone CBT versus AI-CBT. All patients will begin with weekly hour-long telephone counseling, but for patients in the AI-CBT group, those who demonstrate a significant treatment response will be stepped down through less resource-intensive alternatives to hour-long contacts, including: (a) 15 minute contacts with a therapist, and (b) CBT clinician feedback provided via interactive voice response calls (IVR). The AI engine will learn what works best in terms of patients' personally-tailored treatment plan based on daily feedback via IVR about patients' pedometer-measured step counts as well as their CBT skill practice and physical functioning. The AI algorithm the investigators will use is designed to be as efficient as possible, so that the system can learn what works best for a given patient based on the collective experience of other similar patients as well as the individual's own history. The investigator's hypothesis is that AI-CBT will result in pain-related functional outcomes that are no worse (and possibly better) than the standard approach, but by scaling back the intensity of contact that is not resulting in marginal gains in pain control, the AI-CBT approach will be significantly less costly in terms of therapy time. Secondary hypotheses are that AI-CBT will result in greater patient engagement and patient satisfaction. Outcomes will be measured at three and six months post recruitment and will include pain-related interference, treatment satisfaction, and treatment dropout.

ELIGIBILITY:
Inclusion Criteria:

* Back pain-related dx including back and spine conditions and nerve compression and a score of >=4 (indicating moderate pain) on the 0-10 Numerical Rating Scale on at least two separate outpatient encounters in the past year
* At least 1 outpatient visit in last 12 months
* At least moderate pain-related disability as determined by a score of 5+on the Roland Morris Disability Questionnaire
* At least moderate musculoskeletal pain as indicated by a pain score of >=4 on the Numeric Rating Scale
* Pain on at least half the days of the prior 6 months as reported on the Chronic Pain item
* Touch-tone cell or land line phone.

Exclusion Criteria:

* COPD requiring oxygen
* Cancer requiring chemotherapy
* Currently receiving CBT
* Suicidality
* Receiving surgical tx related to back pain
* Active psychotic symptoms
* Severe depressive symptoms
* Can't speak English
* Sensory deficits that would impair participation in telephone calls
* Patient not planning to get care at study site
* PCP not affiliated with study site
* Limited life expectancy (COPD requiring oxygen or Cancer requiring chemotherapy
* Active psychotic symptoms, suicidality, severe depressive symptoms (Beck Depression Inventory (BDI) score or 30+)
* Substance use disorder or dependence, active manic episode, or poorly controlled bipolar disorder as identified by MMini International Neuropsychiatric Interview
* Severe depression identified by chart review of diagnoses and mental health treatment notes
* Cognitive impairment defined by a score of <=5 on the Six-Item screener
* Current CBT or surgical treatment related to back pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Piette, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Alicia A. Heapy, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No
No/Undecided

REFERENCES:
- [Result] Piette JD, Newman S, Krein SL, Marinec N, Chen J, Williams DA, Edmond SN, Driscoll M, LaChappelle KM, Kerns RD, Maly M, Kim HM, Farris KB, Higgins DM, Buta E, Heapy AA. Patient-Centered Pain Care Using Artificial Intelligence and Mobile Health Tools: A Randomized Comparative Effectiveness Trial. JAMA Intern Med. 2022 Sep 1;182(9):975-983. doi: 10.1001/jamainternmed.2022.3178. PMID 35939288
- [Result] MacLean RR, Buta E, Higgins DM, Driscoll MA, Edmond SN, LaChappelle KM, Ankawi B, Krein SL, Piette JD, Heapy AA. Using Daily Ratings to Examine Treatment Dose and Response in Cognitive Behavioral Therapy for Chronic Pain: A Secondary Analysis of the Co-Operative Pain Education and Self-Management Clinical Trial. Pain Med. 2023 Jul 5;24(7):846-854. doi: 10.1093/pm/pnac192. PMID 36484691
- [Result] Mattocks KM, LaChappelle KM, Krein SL, DeBar LL, Martino S, Edmond S, Ankawi B, MacLean RR, Higgins DM, Murphy JL, Cooper E, Heapy AA. Pre-implementation formative evaluation of cooperative pain education and self-management expanding treatment for real-world access: A pragmatic pain trial. Pain Pract. 2023 Apr;23(4):338-348. doi: 10.1111/papr.13195. Epub 2022 Dec 29. PMID 36527287
- [Result] Piette JD, Krein SL, Striplin D, Marinec N, Kerns RD, Farris KB, Singh S, An L, Heapy AA. Patient-Centered Pain Care Using Artificial Intelligence and Mobile Health Tools: Protocol for a Randomized Study Funded by the US Department of Veterans Affairs Health Services Research and Development Program. JMIR Res Protoc. 2016 Apr 7;5(2):e53. doi: 10.2196/resprot.4995. PMID 27056770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AI CBT | Standard Telephone CBT
Started | 166 | 112
Completed | 151 | 100
Not Completed | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AI CBT | Standard Telephone CBT | Total
Number analyzed (Participants) | 166 | 112 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (13.1) | 65.6 (10.6) | 63.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 9 | 30
  Male | 145 | 103 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 160 | 105 | 265
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 10 | 37
  White | 131 | 94 | 225
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 0 | 1 | 1
Pain-related Disability [Mean (Standard Deviation); unit: units on a scale] — The Roland Morris Disability Questionnaire (RMDQ) is a 24-item checklist designed for patients to identify the level of disability and functional status associated with chronic low back pain. Patients are instructed to endorse items that describe their functional status that day. Scores range from 0-24, with higher scores indicating more disability.
  units on a scale | 13.7 (4.1) | 13.5 (4.2) | 13.6 (4.1)
Global Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — An 11-point Numeric Rating Scale (NRS) for pain severity, with 0 representing "No pain" and 10 representing the "Worst pain imaginable." Patients were asked to rate their level of pain on average in the last week.
  units on a scale | 6.2 (1.6) | 6.3 (1.4) | 6.2 (1.5)
Pain-Related Interference [Mean (Standard Deviation); unit: units on a scale] — Pain-related interference was measured using the Brief Pain Inventory - Short Form (BPI). Scores range from 0-10, with higher scores indicating more interference.
  units on a scale | 4.9 (2.2) | 5.0 (2.1) | 4.9 (2.1)
Depression Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Depression symptom severity was assessed using the 9-item Patient Health Questionnaire (PHQ-9). Scores range from 0-27, with higher scores indicating more depression symptom severity.
  units on a scale | 6.3 (5.2) | 6.6 (5.1) | 6.5 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Pain-related Disability
Description: The Roland Morris Disability Questionnaire (RMDQ) is a 24-item checklist designed for patients to identify the level of disability and functional status associated with chronic low back pain. Patients are instructed to endorse items that describe their functional status that day. Scores range from 0-24, with higher scores indicating more disability.
Time Frame: 3 and 6 months post enrollment
Population: The number analyzed in rows differs because some participants did not complete the questionnaire at all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AI CBT | Standard Telephone CBT
Number analyzed (Participants) | 151 | 100
units on a scale
  3 months post enrollment: number analyzed (Participants) | 143 | 92
  3 months post enrollment | 11.0 (6.1) | 11.3 (5.1)
  6 months post enrollment: number analyzed (Participants) | 137 | 97
  6 months post enrollment | 11.0 (5.9) | 12.6 (5.3)

2. Secondary Outcome: Global Pain Intensity
Description: An 11-point Numeric Rating Scale (NRS) for pain severity, with 0 representing "No pain" and 10 representing the "Worst pain imaginable." Patients were asked to rate their level of pain on average in the last week.
Time Frame: 3 and 6 months post enrollment
Population: The number analyzed in rows differs because some participants did not complete the questionnaire at all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AI CBT | Standard Telephone CBT
Number analyzed (Participants) | 151 | 100
units on a scale
  3 months post enrollment: number analyzed (Participants) | 140 | 91
  3 months post enrollment | 5.1 (2.0) | 5.0 (1.8)
  6 months post enrollment: number analyzed (Participants) | 136 | 96
  6 months post enrollment | 5.3 (1.9) | 5.7 (1.9)

3. Secondary Outcome: Pain-Related Interference
Description: Pain-related interference was measured using the Brief Pain Inventory - Short Form (BPI). Scores range from 0-10, with higher scores indicating more interference.
Time Frame: 3 and 6 months post enrollment
Population: The number analyzed in rows differs because some participants did not complete the questionnaire at all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AI CBT | Standard Telephone CBT
Number analyzed (Participants) | 151 | 100
units on a scale
  3 months post enrollment: number analyzed (Participants) | 143 | 91
  3 months post enrollment | 3.9 (2.4) | 3.8 (2.1)
  6 months post enrollment: number analyzed (Participants) | 136 | 95
  6 months post enrollment | 3.9 (2.3) | 4.5 (2.6)

4. Secondary Outcome: Depression Symptom Severity
Description: Depression symptom severity was assessed using the 9-item Patient Health Questionnaire (PHQ-9). Scores range from 0-27, with higher scores indicating more depression symptom severity.
Time Frame: 3 and 6 months post enrollment
Population: The number analyzed in rows differs because some participants did not complete the questionnaire at all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AI CBT | Standard Telephone CBT
Number analyzed (Participants) | 151 | 100
units on a scale
  3 months post enrollment: number analyzed (Participants) | 143 | 92
  3 months post enrollment | 6.7 (5.3) | 6.7 (5.1)
  6 months post enrollment: number analyzed (Participants) | 136 | 96
  6 months post enrollment | 6.8 (5.1) | 7.5 (6.0)

ADVERSE EVENTS:
Time Frame: During the intervention period (approximately 10 weeks of the standard telephone CBT or the AI CBT).
Arm/Group | AI CBT | Standard Telephone CBT
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/112
Serious Adverse Events (participants affected / at risk) | 5/166 | 3/112
Other Adverse Events (participants affected / at risk) | 0/166 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AI CBT (N=166) | Standard Telephone CBT (N=112)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Unrelated to study
Stroke (Vascular disorders) | 1 (1) | 0 (0) — Unrelated to study
Infection (Infections and infestations) | 2 (2) | 1 (1) — Unrelated to study
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated to study
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated to study
Heat stroke (General disorders) | 0 (0) | 1 (1) — Unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT02464449/Prot_SAP_000.pdf